CLINICAL TRIAL: NCT00254332
Title: Effect of Denileukin Diftitox in T-Regulatory Cells in CTCL Patients
Brief Title: Effect of Denileukin Diftitox on Immune System in CTCL Patients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Other Study IDs: IRB 0509084
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2007-12

CONDITIONS: Cutaneous T-cell Lymphoma; Sezary Syndrome; Mycosis Fungoides
Keywords: Cutaneous T-cell Lymphoma; Sezary Syndrome; Mycosis Fungoides; Denileukin Diftitox
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Sezary Syndrome; Mycosis Fungoides

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a blood and tissue study to determine the effect of the drug called denileukin diftitox on the immune system cells that may be involved in patient response to their cutaneous t-cell lymphoma.

Patients who are undergoing standard of care therapy with denileukin diftitox will be invited to participate. Blood and tissue samples will be obtained at baseline, day 5 and day 19 in up to the first 4 cycles of denileukin diftitox.

DETAILED DESCRIPTION:
Although the etiology of CTCL is not fully understood, it is believed to be a malignancy proliferation of a "memory" T-cell in the context of Th2-type cytokine profile and suppressed cytotoxic T-cell (CTL) immunity. T-regulatory (T-regs) cells may be important in CTCL in the setting of immunotherapy. Removal of T-regs would result in enhanced immune responses in vitro, which may translate into augmentation of the anti-tumor immune response and durable clinical responses in vivo. We propose to evaluate effects of ONTAK on the T-reg cell subset in patients undergoing routine therapy with ONTAK. We will evaluate T-reg subsets in peripheral blood and tumor tissues from the patients both phenotypically using multi-color FACS analysis and confocal microscopy, and functionally in MLRs and ELISpot assays with baseline, day 5 and 19 blood samples in up to four cycles.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* diagnosed with CTCL
* able and willing to provide informed consent
* will be receiving denileukin diftitox per standard guidelines

Exclusion Criteria:

* prior history of receiving Ontak
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-11; Study Completion 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Larisa J. Geskin, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsubrgh Medical Center, Pittsburgh, Pennsylvania, United States